CLINICAL TRIAL: NCT07378306
Title: FAsting-mimicking Diet in Combination With Neoadjuvant Chemo-immunoTherapy for Early or Locally Advanced Triple-Negative Breast Cancer: the Prospective, Single-arm, Open-lable, Phase 2 FACT-TN Trial
Brief Title: FMD and Neoadjuvant Chemo-immunotherapy in TNBC
Acronym: FACT-TN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Si-Yu Wang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-861-01; GASTO-10140 (Other: Guangdong Association of Study of Thoracic Oncology)
Record Dates: First submitted 2026-01-16; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: triple-negative breast cancer; fasting-mimicking diet; neoadjuvant; chemo-immunotherapy
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Drug Therapy; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMD plus chemo-immunotherapy (Experimental): The treatment regimen comprises neoadjuvant standard chemotherapy combined with toripalimab, delivered simultaneously with a fasting-mimicking diet intervention.
  Interventions: Other: Fasting-mimicking diet; Drug: Chemotherapy; Drug: Toripalimab

INTERVENTIONS:
Other: Fasting-mimicking diet — The Fasting-Mimicking Diet (FMD) will be administered every three weeks for a maximum of 8 consecutive cycles, unless side effects necessitate its temporary or permanent discontinuation. Each FMD cycle will consist of a specific FMD regimen for five consecutive days, repeated every three weeks.
  The FMD regimen is a plant-based, low-calorie (approximately 738 kcal on Day 1; approximately 536 kcal on Days 2 to 5), low-protein, low-carbohydrate diet. All patients will follow the identical prescribed FMD regimen. No modifications or personalization to the prescribed FMD plan is permitted. The first FMD cycle will commence two days before the administration of the first cycle of chemoimmunotherapy, be applied on the day of chemotherapy, and continue for two additional days after chemotherapy concludes.
  Other Names: FMD
Drug: Chemotherapy — All enrolled patients received standard preoperative chemotherapy combined with anti-PD-1 therapy. The neoadjuvant regimens were guideline-recommended protocols: TP×4-AC×4 combined with PD-1 inhibitor, TP plus PD-1 inhibitor, or PD-1 inhibitor combined with other taxane-based regimens.
  * T: Taxanes, including docetaxel, nab-paclitaxel, and paclitaxel.
  * P: Platinum agents.
  * A: Anthracyclines, including epirubicin, pirarubicin, and doxorubicin.
  * C: Cyclophosphamide.
  Other Names: chemo
Drug: Toripalimab — In the neoadjuvant phase, toripalimab (anti-PD-1) was dosed intravenously at 240 mg on day 1 of every 21-day cycle.
  Other Names: JS001

SUMMARY:
The primary objective of this study is to investigate the efficacy and safety of a fasting-mimicking diet (FMD) intervention combined with standard neoadjuvant chemoimmunotherapy in early-stage or locally advanced triple-negative breast cancer (TNBC).

DETAILED DESCRIPTION:
Despite the significantly superior efficacy of neoadjuvant chemoimmunotherapy, a considerable proportion of early-stage treated triple-negative breast cancer (TNBC) patients ultimately experience recurrence, particularly those who do not achieve pathological complete response (pCR) after surgery. Therefore, there is an urgent need to develop new and effective treatment strategies to improve outcomes for TNBC patients. Additionally, selecting patients who are more likely to benefit from neoadjuvant chemotherapy combined with immunotherapy remains a clinical challenge. The fasting-mimicking diet (FMD) is a strictly calorie-restricted, low-sugar, low-protein, and high-fat dietary regimen that shares metabolic and anti-tumor effects with water-only fasting while reducing the risk of severe adverse reactions, leading to extensive exploration in both preclinical and clinical settings. Numerous clinical trials in breast cancer and various other cancers have investigated FMD, consistently demonstrating that FMD enhances the efficacy of standard anti-tumor therapies with a favorable safety profile. Furthermore, FMD has shown potent immunomodulatory effects in both in vivo studies and cancer patients, with the activation of anti-tumor immunity being a key mechanism underlying the anti-cancer effects of FMD alone or in combination with chemotherapy. Based on the above research background, this study focuses on operable early-stage or locally advanced triple-negative or near-triple-negative breast cancer. Patients will receive neoadjuvant standard chemotherapy combined with immunotherapy alongside FMD dietary intervention, aiming to explore the efficacy and safety of FMD dietary intervention in combination with standard neoadjuvant therapy for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient or their legal representative.
* Good patient compliance, willing and able to adhere to the prescribed dietary intervention plan, visits, treatment schedule, laboratory tests, and other study procedures.
* Female, aged 18 to 70 years.
* ECOG performance status score of 0 to 1, with an expected survival of >12 weeks.
* Female patients of childbearing potential must agree to use reliable methods of contraception from before trial entry, throughout the study, and for 8 weeks after the completion of the study.
* Patients with pathologically confirmed primary breast cancer, with a primary tumor ≥2 cm and regional lymph node status N0-N3 (AJCC Version 8); patients with positive lymph nodes may have a primary tumor of any size; no distant metastases (M0).
* Triple-negative or near-triple-negative subtype, defined as HR-negative or low expression (ER and/or PR positivity rate 1%-10%) and HER2-negative (IHC 0, 1+, or 2+ with FISH-negative).
* No prior history of any anti-tumor therapy, including chemotherapy, radiotherapy, and biological therapy.
* Hemoglobin ≥90 g/L (can be maintained or exceed this level via transfusion).
* Absolute neutrophil count ≥1.5 × 10E9/L.
* Platelet count ≥100 × 10E9/L.
* Total bilirubin ≤1.5 × upper limit of normal (ULN).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN.
* Creatinine ≤1.5 × ULN.
* Fasting blood glucose <250 mg/dL (13.89 mmol/L).
* Pregnancy must be ruled out for women of childbearing potential (aged 15-49).

Exclusion Criteria:

* Previous administration of any systemic anti-cancer therapy, including cytotoxic chemotherapy, targeted therapy, immunotherapy, or investigational treatment.
* Prior radiotherapy for breast cancer.
* Documented evidence (pathological or radiological) of distant metastasis prior to treatment initiation.
* History of another malignancy within the five years preceding treatment initiation in this study, except for carcinoma in situ of the cervix, cured basal cell carcinoma, or urothelial tumors of the bladder (including Ta and Tis).
* Known allergy or hypersensitivity to any component of the investigational drugs or products.
* Active autoimmune disease requiring systemic treatment (e.g., systemic lupus erythematosus, psoriasis, etc.).
* Body Mass Index (BMI) < 19 kg/m².
* Unintentional weight loss ≥5% within the past 3 months, unless the patient's BMI >22 kg/m² and weight loss at study entry is <10%; or unintentional weight loss ≥10% within the past 3 months, unless the patient's BMI >25 kg/m² and weight loss at study entry is <15%. In either case, weight must have been stable for at least one month prior to enrollment.
* Eating disorders, including anorexia nervosa, bulimia nervosa, etc.
* Baseline fasting blood glucose ≤60 mg/dL (3.33 mmol/L).
* Severe infection within 4 weeks prior to enrollment, including but not limited to hospitalization for infectious complications, bacteremia, or severe pneumonia.
* Type 1 or Type 2 diabetes mellitus requiring medication (including but not limited to insulin or insulin secretagogues), with the exception of metformin.
* Any unstable systemic disease, including: uncontrolled hypertension, unstable angina, angina pectoris with onset within the last 3 months, congestive heart failure, myocardial infarction (within 6 months prior to enrollment).
* Severe arrhythmia requiring medication, or significant hepatic, renal, or metabolic disease.
* Known infection with Human Immunodeficiency Virus (HIV).
* Active, uncontrolled hepatitis B or hepatitis C.
* Pregnant or lactating women.
* History of diagnosed neurological or psychiatric disorders, including epilepsy or dementia.
* Any other condition deemed by the investigator as unsuitable for participation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Total pathological complete response (pCR) rate | One week post-operation for the last enrolled patient
  The number of patients with pCR out of the total number of participants using a definition of ypT0/Tis ypN0 after neoadjuvant therapy and surgery.

SECONDARY OUTCOMES:
Rate of Residual Cancer Burden (RCB) of 0-1 | One week post-operation for the last enrolled patient.
  The number of patients with RCB of 0-1 after neoadjuvant therapy and surgery.
Objective Response Rate (ORR) | Two weeks after the end of the final cycle (each cycle is 21 days) for the last enrolled patient.
  The number of patients with complete response and partial response out of the total number of participants
Event-Free Survival (EFS) | Three years after the last patient is enrolled
  EFS was defined as the time from registration to disease progression (local relapse or distant metastases) or death from any cause, whichever came first
Adverse events (AEs) | One year after the last patient is enrolled
  Adverse events (AEs) were graded according to NCI CTCAE v5.0.
Change in Quality of Life (QoL) scores on the EORTC QLQ-C30 questionnaire | From baseline to 3 years after surgery
  Scores obtained on the scales of the EORTC QLQ-C30. Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Change in Quality of Life (QoL) scores on the EORTC QLQ-BR 23 questionnaire | From baseline to 3 years after surgery
  This EORTC breast cancer specific QLQ-BR23 questionnaire is intended to supplement the QLQ-C30.
  The QLQ-BR23 contains 23 items incorporating five multi-item scales to assess systemic therapy side effects, arm symptoms, breast symptoms, body image and sexual functioning. In addition, single items assess sexual enjoyment, hair loss and future perspective. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. For all items but sexual functioning and sexual enjoyment, higher scores indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Tang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Statistical Analysis Plan (SAP) will be shared with other researchers after publication of the study.
Supporting Information: Study Protocol, SAP